CLINICAL TRIAL: NCT03458104
Title: Modeling the Effects of Vocal Cord Atrophy on Airflow and Voice Quality in Elderly Individuals
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment logistics
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Pro00076393
Record Dates: First submitted 2018-02-09; First posted 2018-03-08 (Actual); Last update posted 2020-04-07 (Actual); Status verified 2020-04

CONDITIONS: Vocal Cord Atrophy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vocal Cord Atrophy (Experimental): Quantify changes in aerodynamic and aeroacoustics patterns in patients with vocal cord atrophy (VCA) before and after voice therapy. To evaluate changes, subjects will have Laryngovideostroboscopy, Acoustic/Auerodynamic testing, and Cone Beam CT scans of the larynx before and after voice therapy.
  Interventions: Other: Cone Beam Computed Tomography; Diagnostic Test: Acoustic/Auerodynamic testing; Diagnostic Test: Laryngovideostroboscopy
- Healthy Volunteer (Active Comparator): Develop a validated computational model for assessing normative laryngeal aerodynamic and aeroacoustic patterns in healthy elderly individuals. To assess normal laryngeal aerodynamic and aeroacoustic patterns in this cohort, subjects will subjects will have Laryngovideostroboscopy, Acoustic/Auerodynamic testing, and Cone Beam CT scans of the larynx.
  Interventions: Other: Cone Beam Computed Tomography; Diagnostic Test: Acoustic/Auerodynamic testing; Diagnostic Test: Laryngovideostroboscopy

INTERVENTIONS:
Other: Cone Beam Computed Tomography — Cone Beam CT of the larynx
Diagnostic Test: Acoustic/Auerodynamic testing — Records and displays real-time sound pressure level intensity, intraoral pressure, airflow rate, and fundamental frequency
Diagnostic Test: Laryngovideostroboscopy — Visualization of vocal cords in slow motion. It uses a stroboscopic lamp, which generates regular flashes of light. A flexible tube is inserted in the back of the mouth or through the nose and into the throat. Video pictures are then recorded while patients are making sound.

SUMMARY:
1. The purpose of this study is to develop a validated computational model for assessing normative change in these patterns in patients with vocal cord atrophy before and after voice therapy.
2. This is a prospective study comparing two cohorts - patients with vocal cord atrophy(VCA) (G1) and healthy controls (G2). Subjects with VCA will receive a cone beam computed tomography (CBCT) scan with the standard laryngeal protocol before and after voice therapy. Healthy controls will also receive one cone beam computed tomography (CBCT) scan. Subjects with VCA (G1) will undergo post-therapy scans approximately 4 weeks after completion of voice therapy treatment. Enrolled subjects will also undergo a video stroboscopy and acoustic/aerodynamic testing. Subjects in G1 typically have these procedures performed before and after voice therapy as standard of care. Participants in G2 (healthy controls) will have the video stroboscopy and acoustic/aerodynamic testing just once since they would not otherwise be scheduled to undergo voice therapy. Potential subjects will be between 65 and 80 years of age will be considered for the study if they qualify based on inclusion criteria. Potential subjects will undergo are pre-screening process involving an initial telephone screening.
3. Raw data (measured and calculated) derived from this pilot study will be reported, and no statistical analysis will be performed. Data from specific aim 1 (G2) and specific aim 2 (G1) will be compared using graphical representations such as bar and dot plots. There is a potential for the loss of confidentiality; however, every reasonable effort will be made to limit breaches of privacy and confidentiality. Subjects may directly benefit from this study. In addition, data and conclusions derived from this study may help future patients regarding the effects of vocal therapy on vocal cord atrophy (VCA).

The investigators will recruit up to 12 subjects to account for screen failures. Once 8 eligible subjects are enrolled (4 per group), then enrollment will end.

ELIGIBILITY:
Healthy Subjects Cohort:

Inclusion criteria:

* Between 65 and 80 years of age
* Voice Handicap Index (VHI) questionnaire score of less than 10.
* Little or no dysphonia as assessed by a speech language pathologist from the Duke Voice Care Center
* No contraindications to have a CBCT scan (as assessed per standard clinical practice)

Exclusion criteria:

* Inability to speak, read, write, and understand English
* Inability to provide written consent
* Self-reported or known allergy to Afrin or Tetracaine HCL (or related class of drugs) and unable or willing to complete the laryngovideostroboscopy procedure with it.

Vocal Cord Atrophy Cohort:

Inclusion criteria:

* Between 65 and 80 years of age
* Clinical diagnosis of vocal cord atrophy (VCA)
* Treated for the above condition by a provider at the Duke Head and Neck Surgery & Communication Sciences Clinic
* Elected to undergo voice therapy as standard of care for treatment of VCA

Exclusion criteria:

* Other conditions that affect the voice and would interfere with study measures, as determined by PI
* Inability to speak, read, write, and understand English
* Inability to provide written consent
* Self-reported or known allergy to Afrin or Tetracaine HCL (or related class of drugs) and unable or willing to complete the laryngovideostroboscopy procedure with it.

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-03-28 (Actual); Primary Completion 2020-09 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
Change in acoustic/aerodynamic quantities as measured by the Phonatory Aerodynamic System | Baseline, 12 weeks
  Composite score of vital capacity, mean airflow rate, laryngeal airway resistance, maximum phonation duration, sound pressure level, frequency, aerodynamci dfficiency

SECONDARY OUTCOMES:
Quantify changes in aerodynamic and aeroacoustics patterns in patients with vocal cord atrophy (VCA) before and after voice therapy. | Baseline, 12 weeks
  before and after treatment changes of aerodynamic and aeroacoustic patterns

CONTACTS AND LOCATIONS:
Overall Officials: Dennis Frank-Ito, PhD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No